CLINICAL TRIAL: NCT06996327
Title: The Potential Role of Compounds Derived From Ultra-processed Foods in the Pathogenesis: the UPAD Project
Brief Title: The Potential Role of Compounds Derived From Ultra-processed Foods in the Pathogenesis of Atopic Dermatitis in Pediatric Age
Acronym: UPAD Project
Status: Recruiting | Type: Observational
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Roberto Berni Canani, MD, PhD, Full Professor, Federico II University
Other Study IDs: 163/2024
Record Dates: First submitted 2025-05-21; First posted 2025-05-30 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-05

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pediatric patients with AD: Pediatric patients with a confirmed diagnosis of atopic dermatitis
  Interventions: Other: Evaluation of dietary consumption of UPFs
- Healthy controls: healthy controls matched for age and sex without atopic dermatitis
  Interventions: Other: Evaluation of dietary consumption of UPFs

INTERVENTIONS:
Other: Evaluation of dietary consumption of UPFs — Evaluation of dietary consumption of ultraprocessed foods

SUMMARY:
Atopic dermatitis (AD) is a common chronic inflammatory skin condition, primarily affecting children in urban and high-income areas. Its prevalence has increased significantly over the past 30 years, with up to 20% of children affected, often within their first year of life. AD is characterized by erythematous, scaly, pruritic lesions, xerosis, and frequent atopy, with distinct clinical features in children compared to adults.

The pathophysiology of AD involves skin barrier dysfunction, immune response alterations, and environmental triggers. Genetic factors, particularly mutations in the filaggrin gene, play a significant role in severe AD, leading to increased water loss and skin dehydration. Immunologically, a Th2-predominant response drives inflammation, and environmental exposures, such as air pollutants and irritants, exacerbate the condition.

Recent studies suggest that dietary habits, particularly a high intake of ultra-processed foods (UPFs), may contribute to AD by activating inflammatory pathways. UPFs, rich in advanced glycation end products (AGEs), induce oxidative stress and inflammation, potentially worsening skin damage. This study aims to explore the potential role of UPF-derived compounds, especially AGEs, in the pathogenesis of pediatric AD.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian subjects, both sexes, age: ≥6 months and ≤10 years, with a confirmed diagnosis of atopic dermatitis, and healthy controls matched for age and sex without atopic dermatitis;
* Written informed consent obtained from the participants and/or their parents/legal guardians.

Exclusion Criteria:

* Non-Caucasian ethnicity; age < 6 or > 10 years
* Presence of other chronic conditions: hypereosinophilic syndrome, fungal or viral infections, connective tissue disorders, autoimmune diseases, vasculitis, bullous dermatoses (e.g., pemphigus), drug hypersensitivity reactions, graft-versus-host disease, monogenic disorders (e.g., Marfan syndrome type 2, Hyper-IgE syndrome)
* Presence of scars, nevi, or unusual skin lesions on both forearms
* Absence of written informed consent

Ages: 6 Months to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Caucasian subjects of both sexes, aged ≥6 and ≤10 years, with a diagnosis of atopic dermatitis, and healthy controls matched for age and sex without atopic dermatitis, recruited from the Pediatric Outpatient Clinics of the University Hospital "Federico II".
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-01-10 (Actual); Primary Completion 2025-01-10 (Actual); Study Completion 2026-01-10 (Estimated)

PRIMARY OUTCOMES:
Comparative evaluation of dietary consumption of ultraprocessed foods (UPFs) | First year
  Comparative evaluation of dietary consumption of UPFs in patients aged from 6 months to 10 years diagnosed with AD and in healthy controls matched for age and sex

SECONDARY OUTCOMES:
Comparative evaluation of dietary consumption of dietary advanced glycation end products (AGEs) | First year
  Comparative evaluation of dietary consumption of dietary AGEs in patients aged from 6 months to 10 years diagnosed with AD and in healthy controls matched for age and sex
Assessment of skin AGEs accumulation level | First year
  Evaluation of subcutaneous AGEs concentrations in patients aged from 6 months to 10 years diagnosed with AD and in healthy controls matched for age and sex
Assessment of the effects of AGEs on the expression of tight junction proteins in human keratinocytes | Second year
  Assessment of the effects of AGEs on the expression of tight junction proteins in human keratinocytes, both under basal conditions and after in vitro stimulation with AGEs
Effects of AGEs intake on SCORAD/EASI scores | First year
  Correlation between AGEs intake and Scoring Atopic Dermatitis (SCORAD Score 0 absent - 130 severe) and Eczema Area and Severity Index (EASI Score 0 absent - 72 severe)
Evaluation of transepidermal water loss (TEWL) | First year
  TEWL assessment

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Traslational Medical Science - University of Naples Federico II, Naples, Italy